CLINICAL TRIAL: NCT05684939
Title: Study of the Relation Between the Consumption of Psychoactive Substances and Pain, in Patients Suffering or Surviving From Cancer and Followed in France: Cross-sectional Pilot Study
Brief Title: Relation Between Substance Use and Pain, in Patients Suffering or Surviving From Cancer and Followed in France
Acronym: CAPS
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2022 BALAYSSAC
Record Dates: First submitted 2023-01-04; First posted 2023-01-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2022-12

CONDITIONS: Cancer; Pain; Substance Use
MeSH Terms: conditions — Neoplasms; Pain; Substance-Related Disorders | interventions — Surveys and Questionnaires; Patient Reported Outcome Measures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- cancer patients and cancer survivors: answer to an online questionnaire
  Interventions: Behavioral: Questionnaire (patient reported outcome)

INTERVENTIONS:
Behavioral: Questionnaire (patient reported outcome) — Online self-administered questionnaire exploring substance use, pain, chemotherapy-induced peripheral neuropathy, health-related quality of life, anxiety, depression, social and material deprivation, patients and oncological charactericitcs, and intercurrent pathologies

SUMMARY:
Pain is one of the most prevalent symptoms during and after cancer. Pain can be the consequence of several situations (disease progression, surgery, and anticancer drugs). However, pain can frequently be associated with a substance use disorder (alcohol, tobacco, drugs, and illicit products such as cannabis). The relationship between substance use and pain is known to be complex and interdependent, i.e. pain can reinforce substance use and substance use can promote pain. However, few data in the literature are available on the use of psychoactive substances in relation to pain in the context of cancer (cancer patients and cancer survivors). Moreover, the scientific literature agrees on the fact that these elements are little studied and underestimated in the clinic.

The investigators hypothesize that, in cancer patients or cancer survivors, the prevalence of the use of psychoactive substances would be higher in the presence of pain, and would be associated with its intensity and its impact on the quality Health-Related Living (HRQoL).

The main objective of this study will be to compare, in an adult population of patients suffering from cancer or having had cancer, the prevalence of the consumption of psychoactive substances in painful patients compared to non-painful patients.

DETAILED DESCRIPTION:
Patients will answer to an online questionnaire thanks to associations of cancer patients and social networks, in order to explore their substance use and pain status.

ELIGIBILITY:
Inclusion Criteria:

- Adult patient, male or female, declaring himself as suffering or having suffered from cancer and recruited as such via appropriate communication systems (patient associations, etc.)

Exclusion Criteria:

* Difficulty to understand French language
* Residence outside France (will be verified by the information from the department at the start of the questionnaire)
* Patient close relative
* Protected adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients and cancer survivors recruited thanks to associations of cancer patients and social networks
Sampling Method: Non-Probability Sample
Enrollment: 2010 (Actual)
Dates: Start 2023-01-27 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
substance use | day 1
  Legal: alcohol, tobacco, electronic cigarette, psychotropic drugs (benzodiazepines, z-drugs, and opioids), CBD, and other susbtances Illegal: cannabis, and other drugs
  At least once in the past year, at least once in the past month, at least once in the past week, or at least once a day

SECONDARY OUTCOMES:
Pain severity | day 1
  Brief pain inventory
Neuropathic pain | day 1
  DN4 interview questionnaire
Analgesic use | day 1
  Ongoing analgesic drugs
Chemotherapy-induced peripheral neuropathy | day 1
  QLQ-CIPN20 questionnaire
Health-related quality of life and symptoms | day 1
  QLQ-C30 questionnaire
Anxiety and depression | day 1
  HADS questionnaire
Material and social deprivation | day 1
  EPICES questionnaire
Sociodemographic characteristics of patient | day 1
  age, sex, height, weight, body mass index, area of residence (urban or rural), socio-professional status (INSEE), and department
Oncological characteristic | day 1
  type of cancer, date of cancer diagnosis, and type of treatment (received and/or ongoing)
Intercurrent pathologies | day 1
  open question

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No